CLINICAL TRIAL: NCT00509028
Title: An Open-label, Multi-center, Long Term Study to Investigate the Safety and Efficacy of Budesonide Turbuhaler® Treatment for 48 Weeks (Following 6 Weeks Phase III Study) in Japanese Children With Bronchial Asthma Aged 5 Years to 15 Years Old
Brief Title: Safety and Efficacy Study of Budesonide (Pulmicort®) Turbuhaler® in Japanese Children With Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5254C00006
Record Dates: First submitted 2007-07-17; First posted 2007-07-31 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Asthma; Bronchial
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BUD - Budesonide (Experimental): Budesonide Turbuhaler 100 mcg (Pulmicort® Turbuhaler®), 100 - 400 mcg daily
  Interventions: Drug: Budesonide
- CONV - Conventional Asthma Therapy (Active Comparator): Conventional Asthma Therapy - according to the Japanese Paediatric Guideline for the Treatment and Management of Asthma and at daily dose as judged by the investigator.
  Interventions: Drug: Conventional Asthma Therapy

INTERVENTIONS:
Drug: Budesonide — Budesonide Turbuhaler 100 mcg (Pulmicort® Turbuhaler®), 100 - 400 mcg daily
  Other Names: Pulmicort® Turbuhaler®
  Arms: BUD - Budesonide
Drug: Conventional Asthma Therapy — According to the Japanese Paediatric Guideline for the Treatment and Management of Asthma and at daily dose as judged by the investigator.
  Arms: CONV - Conventional Asthma Therapy

SUMMARY:
This study will include the patients who are Japanese children with bronchial asthma aged 5 years to 15 years old and have completed the Phase III study (Study code: D5254C00769) at about 29 centres. To investigate the safety of budesonide Turbuhaler® with a daily dose of 100 µg to 800 µg for 54 weeks treatment including the prior 6 weeks Phase III study (Study D5254C00769, NCT00504062) as compared with conventional therapy in Japanese children with bronchial asthma in need of inhaled glucocorticosteroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who complete preceding the Phase III study and provide a signed written informed consent by patient's legal representative at Visit 1 or 4 weeks prior to Visit 1 of the study. A signed written informed assent should also be obtained from the patients themselves as much as possible
* When the investigator will obtain the signed written informed consent of Phase III study (D5254C00769) from patient's legal representative, the investigator will also provide the information of this study

Exclusion Criteria:

* Respiratory infections that, in the opinion of the investigator(s), may affect the efficacy evaluation e.g., lower airways infection such as pneumonia, infection with no available effective antimicrobial drugs or with deep seated mycosis
* Concurrent serious diseases of liver, kidney, heart or other complications which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study. Any clinically relevant abnormal findings in vital sign or physical examination at Visit 1 in this study, which in the opinion of the investigator may put the patient at risk because of his/her participation in the study.
* Pregnant or possible pregnancy or planning to become pregnant during the study period
* Other subjects who are considered inappropriate to participate in this study judged by the investigator

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Goran Carlsson, MD, Study Director — AstraZeneca R&D Lund
Locations (1):
- Research Site, Takizawa, Iwate, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 241 Japanese paediatric patients were enrolled into the study
Pre-assignment Details: This was an open-label, multi-centre, long-term study in Japanese children with bronchial asthma aged 5 to 15 years, and conducted as an extension of the Phase III study D5254C00769.
Groups:
- Conventional Therapy: According to the Japanese Paediatric Guideline for the Treatment and Management of Asthma and at daily dose as judged by the investigator.
Period: Overall Study
Arm/Group | Budesonide | Conventional Therapy
Started | 121 | 120
Completed | 109 | 113
Not Completed | 12 | 7
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Non-compliance | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide | Conventional Therapy | Total
Number analyzed (Participants) | 121 | 120 | 241
Age Continuous [Mean (Standard Deviation); unit: Years] | 8.9 (2.6) | 8.6 (2.3) | 8.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 27 | 63
  Male | 85 | 93 | 178

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs).
Description: AEs were defined as undesirable medical conditions or deteriorations of a pre-existing medical condition following/during exposure. All Serious AEs, AEs leading to withdrawal, Other relevant AE were recorded.
Time Frame: 54 weeks
Measure: Number; unit: Participants
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 120
Participants | 118 | 116

2. Secondary Outcome: Number of Patients With Abnormal Clinical Laboratory Test Values.
Description: Analysis of haematological, clinical chemistry and urynalysis variables were performed.
  Haematology variables: erythrocytes, haemoglobin, haematocrit, leucocyte count, leucocyte different count (neutrophils, eosinophils, basophils, lymphocytes, monocytes), platelet count.
  Clinical chemistry measurements: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin, albumin, creatinine,sodium, potassium, total protein, blood urea nitrogen.
  Urinalysis variables: protein, glucose, urobilinogen, occult.
Time Frame: 54 weeks
Measure: Number; unit: Participants
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 120
Participants | 0 | 0

3. Secondary Outcome: Number of Patients With Abnormal Vital Sign Values for the Following Variables: Blood Pressure (Sitting) and Pulse Rate (Sitting), as Judged by the Investigator
Time Frame: 54 weeks
Measure: Number; unit: Participants
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 120
Participants | 0 | 0

4. Secondary Outcome: Number of Patients With Abnormal Plasma Cortisol Values.
Description: Cut-off value of cortisol is defined as 4 mcg/dL.
Time Frame: 54 weeks
Measure: Number; unit: Participants
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 120
Participants | 20 | 12

5. Secondary Outcome: Height
Description: Height, change from baseline calculated as (height at last visit - height at randomization)
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 109 | 113
Centimeters | 5.34 (1.99) | 6.35 (1.89)

6. Secondary Outcome: Weight
Description: Weight, change from baseline calculated as (weight at last visit - weight at randomization)
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 109 | 113
kilograms | 3.78 (2.77) | 4.39 (3.22)

7. Secondary Outcome: Morning Peak Expiratory Flow (PEF) Percentage of Predicted Normal
Description: Change in PEF percent of predicted normal calculated as (PEF percent predicted normal at last visit - PEF percent predicted normal at randomization).
Time Frame: 54 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 120
Percentage | 9.54 (19.87) | 5.84 (17.81)

8. Secondary Outcome: Change From Baseline of Respiratory Condition at Asthma Attacks (Daytime)
Description: Change in respiratory condition at asthma attacks (daytime) from baseline to last visit. Scale: 0 - 4.
  0 = None. 1 = Mild. 2 = Moderate. 3= Severe. 4 = Respiratory insufficiency
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 119
Points on a scale | -0.139 (0.334) | -0.156 (0.302)

9. Secondary Outcome: Change From Baseline of Respiratory Condition at Asthma Attacks (Nighttime)
Description: Change in respiratory condition at asthma attacks (nighttime) from baseline calculated as (respiratory condition at asthma attacks (nighttime) at last visit - respiratory condition at asthma attacks (night-time) at randomization).
  Scale: 0 - 4. 0 = None. 1 = Mild. 2 = Moderate. 3= Severe. 4 = Respiratory insufficiency.
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 119
Points on a scale | -0.12 (0.29) | -0.147 (0.3)

10. Secondary Outcome: Change From Baseline of Use of Inhaled Short-acting B-2 Agonist (Daytime)
Description: Change in use of inhaled short-acting B-2 agonist (daytime) from baseline calculated as (use of inhaled short-acting B-2 agonist (daytime) at last visit - use of inhaled short-acting B-2 agonist (daytime) at randomization)
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Puffs per day
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 119
Puffs per day | -0.21 (0.647) | -0.242 (0.485)

11. Secondary Outcome: Change From Baseline of Use of Inhaled Short-acting B-2 Agonist (Night-time)
Description: Change in use of inhaled short-acting B-2 agonist (night-time) from baseline calculated as (use of inhaled short-acting B-2 agonist (night-time) at last visit - use of inhaled short-acting B-2 agonist (night-time) at randomization)
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Puffs per day
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 119
Puffs per day | -0.07 (0.415) | -0.097 (0.368)

12. Secondary Outcome: Change From Baseline in Disturbance of Daily Activities
Description: Change in disturbance of daily activities from baseline calculated as (disturbance of daily activities at last visit - disturbance of daily activities at randomization).
  Frequency of disturbance of daily activity was assessed using 3- grade scale (normal, almost able, unable).
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Disturbances per day
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 119
Disturbances per day | -0.037 (0.141) | -0.017 (0.141)

13. Secondary Outcome: Change From Baseline in Disturbance of Night-time Sleep
Description: Change in disturbance of night-time sleep from baseline calculated as (disturbances of night-time sleep at last visit - disturbances of night-time sleep at randomization).
  Frequency of disturbance of night- time sleep was assessed using 3- grade scale (normal, almost able, unable).
Time Frame: Baseline and 54 weeks
Measure: Mean (Standard Deviation); unit: Disturbances per night
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 119
Disturbances per night | -0.029 (0.134) | -0.042 (0.132)

14. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Percentage of Predicted Normal Change From Baseline
Description: Forced Expiratory Volume in one second (FEV1) percentage of predicted normal change from baseline calculated as: 100 * (FEV1 at last visit - FEV1 at randomization)/predicted normal FEV1).
Time Frame: 54 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Budesonide | Conventional Therapy
Number analyzed (Participants) | 121 | 120
Percentage | 1.5 (15.59) | 2.31 (16.63)

ADVERSE EVENTS:
Arm/Group | Budesonide | Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 10/121 | 11/120
Other Adverse Events (participants affected / at risk) | 100/121 | 113/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide (N=121) | Conventional Therapy (N=120)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide (N=121) | Conventional Therapy (N=120)
Conjunctivitis Allergic (Eye disorders) | 15 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 68 | 60
Bronchitis (Infections and infestations) | 40 | 46
Pharyngitis (Infections and infestations) | 36 | 40
Gastroenteritis (Infections and infestations) | 28 | 30
Influenza (Infections and infestations) | 30 | 27
Nasopharyngitis (Infections and infestations) | 23 | 21
Otitis Media (Infections and infestations) | 15 | 15
Chronic Sinusitis (Infections and infestations) | 14 | 10
Acute Tonsillitis (Infections and infestations) | 10 | 9
Impetigo (Infections and infestations) | 8 | 9
Hordeolum (Infections and infestations) | 0 | 6
Contusion (Injury, poisoning and procedural complications) | 8 | 9
Headache (Nervous system disorders) | 10 | 11
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 26 | 22
Eczema (Skin and subcutaneous tissue disorders) | 11 | 16
Urticaria (Skin and subcutaneous tissue disorders) | 10 | 12
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 6 | 6
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 6
Heat Rash (Skin and subcutaneous tissue disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less